

| EPD D7 | EPD D700 Protocol | |
|--------------|-------------------|---------|
| Document No. | Revision: | Page |
| CLN-D700-004 | 2.0 | 1 of 15 |

# **DURABLE-I STUDY PROTOCOL** SIGNATURE PAGE

| AUTHORIZATION | | | |
|---|---|---|---|
| | NAME | SIGNATURE | DATE |
| Issued by: | Yitzhack Schwartz, MD<br>Chief Medical Director | V . Schwark | 18.9.2016 |
| Approved | Itzik Shmaayahoo,<br>Director of System<br>Architecture & SW | A CONTRACTOR OF THE PARTY OF TH | 18 0.2 16 |
| by: | Micha Nisani,<br>General Manager | of the si | 18.9.2016 |
| | ment was | Philociline | |

| REVISION HI<br>Revision | | |
|-------------------------|-----------------------------------|------------|
| # | UE scription | Date |
| 1 | First Issue | 14/09/2016 |
| 2 | Up ner. follow, as general Periar | 18.9.2016 |
| | S M | |
| | 11/2 | |
| | 76 40. | |
| Cleur | O. Virginia | |
| (0) | | |
| <b>40</b> | | |
| | | MACTED |
| | | MATER |

MASTER



#### **EPD D700 Protocol**

Document No. CLN-D700-004

Revision: **2.0** 

Page **2 of 15** 

#### **DURABLE-I STUDY:**

#### DIELECTRIC UNRAVELLING OF RADIOFREQUENCY ABLATION EFFECTIVENESS

#### **Study Purpose**

The purpose of this study is to evaluate real-time gap detection using EPD D700 dielectric sensing compared with customary electrical isolation tests and Adenosine infusion at the end of the procedure. Furthermore, safety, usability and clinical applicability of the system for guided AF ablatical be confirmed.

## **Study Design**

Prospective, single-center, non-randomized, non-blinded, open label, and single arm study.

All procedures will be performed under CARTO 3 guidators for the deatment of atrial fibrillation (AF). The EPD 0.700 system will be used interchangably, to record pre-, during and immediate post-ablation tissue character of cs and compute likelihood of lesion transmurality and permanency. Additionally, D700 system safety, feasibility, usability and direct applicability will be obcumented.

The entire procedure will be conducted as customary, using standard and approved off the shelf equipment (body surface electrodes, diagnostic and irrigated ablotion cathete's, RF generator and recording system), in a completely clinically excependent manner from the EPD D700 system. The physician will neither use nor rely on any of the D700 system output for clinical decision making and will be blinded to the D700 lesion assessment forecasts. One month following the initial procedure, a repeated of occurrence will be performed for gap detection and its results will be correlated with the D700 predictions.

# Study Population

Twenty tour Parocysmal Atrial-Fibrillation (PAF) patients, amenable to catheter-basic AF ablation therapy comprising of Pulmonary Veins Isolation (PVI). We suggest that 4 will patients decline to participate. The overall number of patients in the study is twenty.

## **Key Inclusion Criteria**

- 1. Male or female patients, age  $\geq$  18 and  $\leq$  80 years.
- Paroxysmal atrial fibrillation (PAF)



| | EPD D7 | 700 Protocol | |
|---|---|---|---|
| <b>DEPD</b> | Document No. CLN-D700-004 | Revision:<br>2.0 | Page<br><b>3 of 15</b> |

- 3. Able to provide written informed consent form to participate in the study, prior to any study related procedures.
- 4. Able and willing to comply with the study protocol requirements.
- 5. A female subject is eligible if not of child bearing potential or has a negative pregnancy test within the previous 7 days.

# **Key Exclusion Criteria**

- 1. Any planned surgical or endovascular intervention within 30 days before or after the index procedures.
- 2. Subject is enrolled in another drug or device study protocol that has not reached its primary endpoint.
- 3. Previous AF ablation therapy.
- 4. Clinical evidence of active coronary ischemia, significant Valvular heart disease, or hemodynamically significant congenical cardiac community.
- 5. Patient had experienced myocardial inforction (MI), stroke (CVA) or transient ischemic attack (T 4) or other new ological dicturbances.
- 6. Patient has a Lacemaker.
- 7. Thrombi detected in the heart.
- 8. Life capactancy loss than 12 months.
- 9. knr wn sevole renal insufficiency.
- 10. Known allergy to Incine.

#### Baseline Assessment

- Eligibility according to inclusion and exclusion criteria.
- Obtaining signed mormed Consent Form (ICF).
- Demographics.
- 1edical history.
- Concomitant medications.
- Disease oriented physical examination including vital signs.
- 12 lead ECG.
- Standard laboratory tests;
  - Complete blood count
  - Coagulation studies if appropriate
  - Serum creatinine and electrolytes
  - Liver function tests
  - CRP
- TTE or TEE.
- Pregnancy test, if applicable.

MASTER

| | EPD D7 | 700 Protocol | |
|-----|--------------|--------------|---------|
| EPD | Document No. | Revision: | Page |
| LID | CLN-D700-004 | 2.0 | 4 of 15 |

#### Study procedures

- Cardiac CT (pre-procedure imaging) or MR.
- CT/MR post-processing and analysis at EPD Research (Caesarea, Israel):
  - Cardiac chambers' segmentation
  - o Electrical fields computation
  - Optional recommended PVI ablation lines
  - Optional preliminary lesion forecast at the point 'evel
- Forwarding the ready to use pre-planned data to the site.
- First AF ablation procedure (Figure 1):
  - o EPD D700 system installed in the EP cath-lab.
  - O Deployment of body surface electrodes (patches) by the ocal EP technician/nurse under supervision of EPD Research fear members, to be used later by both the School and EPD D700 system, interchangeably, according to the diagrams in Appendix 1.
  - Deployment of BWI booy surface magnetic serious according to the customary setup generalines
  - o Connecting the The moCool smartTouch ablation excheter via the commercially available recension cross to the LARIO3 system according to the diagrams in Appendix 1.
  - O Connecting the Scockert RF abilition generator to the CARTO3 system according to the diagrams in Appendix 1.
  - O Registration of the pre-actuared 3.7 °T or MR images of the Right Arium (3.1) vith EPD D 700, using OrtoMERGE module.
  - Registration of the ore-acquired 3D CT or MR images of the RA with EPD D700 systom under fluoroscopy and or CARTO3-guidance.
  - O Performance of Transsectal Procedure under fluoroscopy and/or ultrasound (TEE or IC.) Buildance.
  - O Registration of the p.e-acquired 3D CT or MR images of the Left At. u.m (LA) and Fulmonary Veins (PVs) with CARTO3 using CARTOMERGE module.
  - Registration of the pre-acquired 3D CT or MR images of the LA and PVs with EPD D700 system under fluoroscopy or CARTO3-guidance.
  - Targeted navigation inside the LA and reaching the 1<sup>st</sup>, either userdetermined or computer recommended, point of the 1<sup>st</sup> preplanned PVI ablation lines.
  - Performing the specific ablation strategy while ascertaining contiguity using VISITAG module, i.e. 5-6 mm between consecutive ablation points, and moving along the PVI line systematically in preplanned continuous order. The specific ablation parameters to be used, i.e. 30 W 30 and 25W a30 sec in anterior and posterior LA wall, respectively; as well as the desired Ablation Index to be reached, will be determined solely by the operator regardless of the system's recommendation.



| | EPD D7 | 700 Protocol | |
|---|---|---|---|
| <b>PEPD</b> | Document No. CLN-D700-004 | Revision:<br>2.0 | Page <b>5 of 15</b> |

- Defore, during and immediately after each ablation point, the EPD D700 system will record (for a few seconds) specific dielectric characteristics from the catheter tip. These readings, reflecting estimated transmurality and probability of the lesion's permanency, will be analyzed in the post-procedure phase and will not be considered by the user during the procedure.
- Thirty minutes after the completion of the full ablation plan, a formal acute electrical isolation test will be performed to identify remaining gaps.
- o IV Adenosine infusion, a bolus of 12-18mg, will be performed to identify additional existing dormant conduction.
- Touch-up ablations will be added according to the two previous tests' findings.
- The procedure will be concluded only after the physician has decided there are currently no remaining identifiable gaps and the PVI is based on current knowledge, deemed durable.



Figure 1: Step-by-step 1st procedure, using both CARTO3 and D700 interchangeably.

## Second AF ablation procedure (Figure 2):

- O The second procedure will be conducted 1 month after the initial procedure in a similar set up under CARTO3 guidance.
- After repeated registration, with the previous pre-acquired 3D image, the LA will be remapped.
- In order to functionally identify existing gaps, remaining gaps will be sought for by electrical functional test.



| | EPD D7 | 700 Protocol | - |
|------------|--------------|--------------|----------------|
| <b>EPD</b> | Document No. | Revision: | Page |
| | CLN-D700-004 | 2.0 | <b>6 of 15</b> |

- If such gaps will be encountered, the physician will apply the customary touch-up approach.
- The location of gaps around the PVs will be reported in 8-16 segments (Figure 3).

## DURABLE - I, 2<sup>nd</sup> Procedure



Figure 2: S'ep-by-s'ep 2nd pro accure, gao de ection and re-isolation.



Figure 3: **Data collection around PVs**. (A) Data collection at 8 numbered sections: 1,9 – superior; 2, 16 – anterior superior; 3, 15 – anterior middle; 4, 14 – anterior inferior; 5, 13 – inferior; 6, 12 – posterior inferior; 7, 11 – posterior middle; 8, 10 – posterior

| | EPD D7 | 00 Protocol | |
|------------|--------------|-------------|----------------|
| <b>EPD</b> | Document No. | Revision: | Page |
| | CLN-D700-004 | 2.0 | <b>7 of 15</b> |

superior; (B) Sections 2, 3, 4 and 14, 15, 16 were grouped, respectively, into left and right anterior segments and 6, 7, 8 and 10, 11, 12 were grouped, respectively, into left and right posterior segments.

# Data to be collected during the procedures:

- Overall procedure time.
- Overall EPD D700 set up time.
- Fluoroscopy time.
- Acute (during and immediately after the procedure) AE/SAE Evaluation

- Lieta Post-ablation

  Lion will be tagged on both

  Is used Contact force data will also be stem data. Pre-ablation, during and Immediat Prost-ablation lesion assessment at each
  - Each ablation site location will be tagged on bot'r ARTO3 and EPD D700
  - As SmartTouch® is used, ontact force data will also be regarded.



| | EPD D | 700 Protocol | |
|---|---|---|---|
| <b>EPD</b> | Document No. CLN-D700-004 | Revision:<br>2.0 | Page <b>8 of 15</b> |

## Appendix 1: CARTO3 and EPD D700 operating in-tandem

This appendix describes the connection between D700 system and CARTO3 (Biosense Webster JNJ) system that was especially developed in order to enable temporary operation of the two systems in-tandem. This is a requirement that must be met merely in the interim phase until users gain full confidence in D700's accuracy and reliability. The connection between the two systems is accomplished by two EPD external boxes:

- EPD CARTO3 Cat box
- EPD CARTO3 Patch box

There are two operational modes enabled while using these connection boxes.

- a. CARTO3 mode:
  - In this mode the CARTO3 is connected as ston lalone system and receins all its customary functionalities using both EM or d Impedance-based localization.
- b. D700 mode:

In this mode the system toggles the F.F. generator and the body surface patches to the D700 system, while disconnecting the CRTO3 from the ablation catheter and the body surface patches. During loads are connected to CARTO3 system as inpute. In this pode, although an error massage might appear on CARTO screen, the CARTO3 is still using its magnitic location and the navigable catheters equipped with a magnetic sensor will still be visualized.

## D700 and Carro3 connection Top level

Figure 1 shows the connection between the two systems.

The control cable carties voltage and control signals for the internal relay box. The connection is made by the two connection boxes:

#### EPD Cart3 Cat box

The EPD Cart3 Cet box is used to connect between the ablation catheter, RF generator, and the D700 system.

Figure 2 shows the internal connections when the box is set to CARTO3 standalone mode. In CARTO3 standalone mode the RF generator is connected directly to CARTO3 and the ablation cacheter electrodes C4-C1 are connected directly to CARTO3. The relay position is set by a control signal from D700. All the relays are hi-voltage enabled and defibrillation safe.

Egure 3 shows the box in the D700 mode. The 13 KHz block filter is used to block the location signals of the D700 from for RF generator low impedance output.

Dummy resistors load are connected to CARTO3 inputs.

#### **EPD Cart3 Patch box**

The EPD Cart3 patches box is used to connect between the body surface patches to CARTO3 or D700 system, interchangeably.



| | EPD D700 Protocol | | |
|---|---|---|---|
| <b>EPD</b> | Document No. CLN-D700-004 | Revision:<br>2.0 | Page <b>9 of 15</b> |

Figure 4 shows the internal connections when the box is set to CARTO3 mode. Figure 5 shows the connection when the box is set to D700 mode.

## **Available Modes**

| CARTOS OTTY | The CARTO3 is connected to all catheter electrodes, body surface patches, and RF generator | Same full performance as standalone CARTO3 system, all indvalling catheters, including SmartTouch |
|---|---|---|
| | surface patches, and RF | all in dv alling catheters, including SmartTouch |
| | TO A CONTROL OF THE STATE OF TH | including SmartTouch |
| 1 | generator | |
| | . 3 | la ation anthotes lane cal |
| | | abiation catheter, Lasso and |
| | | Decapolar diagnost'c |
| | _0 | catheters, and all their |
| | × | electrodes will Lo visualized |
| | | on the CAR O screen |
| D/00 . | 1. | <ul> <li>No RF performance</li> </ul> |
| CARTO3 in EM location only | The CARTO? is connected only | degradat or (energy |
| | to electromagnetic an 1 | transfer) in C1. |
| | tempciature sersois, lence | <ul> <li>ECG_ignals of C1 to</li> </ul> |
| 3 | the abiation catheter will stul | €4 transferred to |
| The state of the s | be correctly localized and | recording system |
| _ | aisplayed or the CARTO | from D700 RS |
| | screen | connection box. |
| | 2. | <ul> <li>Error message on</li> </ul> |
| | Atlation catheter C4-C1 | CARTO screen due to |
| | connected to り700, CA n ている is | "loss" of impedance |
| 20 5 | optionally connected to | input. |
| 0 | dumminoad | <ul> <li>Non-navigation</li> </ul> |
| .6 | 3.0 | diagnostic catheters, |
| | RF general : is connected to | whose visualization |
| .6 | C1 with a blocking filter of | solely depends on |
| | D700 frequencies | impedance |
| | 4. | measurements (body |
| .01 | Body surface patches are | surface patches |
| 20 20 | connected to D700 | reading the current |
| 0, 7/2 | 5. | injected from the |
| | CARTO3 body surface input is | electrodes on the |
| .0) | optionally connected to | catheter), will |
| | dummy load | temporarily |
| | | disappear from the |
| | | CARTO screen |
| | | <ul> <li>The intra-cardiac</li> </ul> |
| | | ECG will be displayed |
| | | on the recording |
| | | system in the |
| | | channels reserved |
| | | for D700 rather than |
| | | the channels |

| EPD D7 | 700 Protocol | |
|--------------|--------------|----------|
| Document No. | Revision: | Page |
| CLN-D700-004 | 2.0 | 10 of 15 |
| | Document No. | |

#### Supported catheters

#### CARTO®3

- 1. NAVISTAR catheter / THERMOCOOL® SF catheter
- 2. THERMOCOOL SMARTTOUCH® catheter 🗸

- 1. CR3425CT 3 m Cable for existing NAV'sTAR® Catheter 25 pin black is in red
  - 2. CR3434CT 3 m Cable fc. THERMOCOO. SMARTTOUCH® Catheter, 24 pin red, 34 pin red















MASTER



| FPD | D700 | Protocol |
|-----|------|----------|

Document No. CLN-D700-004

Revision: 2.0

Page **14 of 15** 







Solid FULL TOOLS BE THE Product at Solid Fruit Tools Base the Country of the Coun